CLINICAL TRIAL: NCT05903768
Title: Comparison of Capsular Stretching and Passive Joint Mobilization in Idiopathic Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah IU Maria Safdar
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Adhesive Capsulitis
Keywords: Range of motion; Shoulder; Pain
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyriax capsular stretching (Experimental): Patient will be subjected to Hot Pack prior to treatment. Detailed intervention will include Active range of motion exercises,Home plan exercises.Anterior, Posterior and inferior capsular stretching.
  Interventions: Other: Cyriax capsular stretching
- Mobilization (Active Comparator): Patient will be subjected to Hot Pack prior to treatment. Detailed intervention will include Active range of motion exercises,Home plan exercises and Maitland's Mobilization:
  Interventions: Other: Mobilization

INTERVENTIONS:
Other: Mobilization — Hot Pack for 5mins,Active range of motion exercises (10 reps x 3 sets),Home plan include: wand exercises, wall-walking exercises, pendulum exercises,towel stretch exercises, Cross Body Adduction (10reps x 2 sets, each)Cold pack for 5 mins.
  Maitland's Mobilization: Inferior glide (10x3), posterior glide, (10 reps x 3 sets), anterior glide (10 reps x 3 sets)
  Arms: Mobilization
Other: Cyriax capsular stretching — Hot Pack for 5mins,Active range of motion exercises (10 reps x 3 sets),Home plan include: wand exercises, wall-walking exercises, pendulum exercises,towel stretch exercises, Cross Body Adduction (10reps x 2 sets, each)Cold pack for 5 mins.
  Anterior, Posterior and inferior capsular stretching would be performed. Each stretch should be held15-30 seconds and repeated 2 to 4 times.
  Arms: Cyriax capsular stretching

SUMMARY:
The aim of this research is to determine the effects of capsular stretching versus passive joint mobilization on Pain, range of motion and Quality of life in patients with Idiopathic Adhesive capsulitis.

DETAILED DESCRIPTION:
In reference study, patients with Adhesive capsulitis were given the option to examine the immediate effects of posterior capsule stretching and scapular mobilization. They came to the conclusion that extending the posterior capsule improved shoulder range of motion. Current study will assess all shoulder movements and also showing effect on Quality of life of patients with adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

Both genders

* Age : 30-50 years
* Pain and Restricted movements of shoulder.
* Patient With Adhesive Capsulitis of Stage 2

Exclusion Criteria:

* Patient with any Intrinsic Etiology such as Haemarthrosis, rheumatoid arthritis ,infection or gout
* Patient with any severe trauma, Shoulder dislocation, subluxation or ligament injury of the shoulder
* Fractures of the shoulder
* Peripheral neurological involvement in the upper extremity.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain rating scale | 4th week
  The Numeric Pain rating scale is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
Range of motion (shoulder flexion) | 4th week
  changes in shoulder flexion Range of motion from baseline to final session was measured
Range of motion (shoulder extension) | 4th week
  changes in shoulder extension Range of motion from baseline to final session was measured
Range of motion (shoulder abduction) | 4th week
  changes in shoulder abduction Range of motion from baseline to final session was measured
Range of motion (shoulder external rotation) | 4th week
  changes in shoulder external rotation Range of motion from baseline to final session was measured
Range of motion (internal rotation) | 4th week
  changes in shoulder internal rotation Range of motion from baseline to final session was measured

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Lady reading hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eckert AJ, Plaumann M, Pehlke S, Beck C, Muhldorfer S, Weickert U, Laimer M, Pfeifer M, Stechemesser L, Holl R. Idiopathic Frozen Shoulder in Individuals with Diabetes: Association with Metabolic Control, Obesity, Antidiabetic Treatment and Demographic Characteristics in Adults with Type 1 or 2 Diabetes from the DPV Registry. Exp Clin Endocrinol Diabetes. 2022 Jul;130(7):468-474. doi: 10.1055/a-1543-8559. Epub 2021 Aug 23. PMID 34425597
- [Background] Thomas SJ, McDougall C, Brown ID, Jaberoo MC, Stearns A, Ashraf R, Fisher M, Kelly IG. Prevalence of symptoms and signs of shoulder problems in people with diabetes mellitus. J Shoulder Elbow Surg. 2007 Nov-Dec;16(6):748-51. doi: 10.1016/j.jse.2007.02.133. PMID 18061115
- [Background] Mengiardi B, Pfirrmann CW, Gerber C, Hodler J, Zanetti M. Frozen shoulder: MR arthrographic findings. Radiology. 2004 Nov;233(2):486-92. doi: 10.1148/radiol.2332031219. Epub 2004 Sep 9. PMID 15358849
- [Background] Janela D, Costa F, Molinos M, Moulder RG, Lains J, Francisco GE, Bento V, Cohen SP, Correia FD. Asynchronous and Tailored Digital Rehabilitation of Chronic Shoulder Pain: A Prospective Longitudinal Cohort Study. J Pain Res. 2022 Jan 8;15:53-66. doi: 10.2147/JPR.S343308. eCollection 2022. PMID 35035234
- [Background] Paul A, Rajkumar JS, Peter S, Lambert L. Effectiveness of sustained stretching of the inferior capsule in the management of a frozen shoulder. Clin Orthop Relat Res. 2014 Jul;472(7):2262-8. doi: 10.1007/s11999-014-3581-2. Epub 2014 Mar 25. PMID 24664198